CLINICAL TRIAL: NCT07346768
Title: Ultrasound Assessment of Anterior Neck Soft Tissue Thickness to Predict Difficult Airway Risk in Obese Patients Undergoing for Surgery Under General Anesthesia: an Observational Study
Brief Title: Evaluation of Anterior Neck Ultrasound in Predicting Difficult Airway in Obese Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Gaziantep City Hospital (Other)
Responsible Party: Principal Investigator, Gamze Nur Teke, Principal Investigator, Gaziantep City Hospital
Other Study IDs: GaziantepCH
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Ultrasonography; Airway Management; Intubation, Intratracheal; Obesity and Overweight
Keywords: Obesity; difficult airway; anterior neck ultrasound; ultrasonography
MeSH Terms: conditions — Obesity; Overweight | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overweight and Obese Surgical Patients: Adult overweight and obese patients undergoing elective surgery under general anesthesia who will receive standard care airway management.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — one group, there is no intervention. All measurements and observations will be performed during routine clinical care only

SUMMARY:
Obese patients are at increased risk of difficult airway management due to anatomical changes in the anterior neck soft tissues. Accurate preoperative prediction of difficult airway remains challenging using conventional clinical airway assessment tests alone.

This prospective observational study aims to evaluate the role of ultrasound assessment of anterior neck soft tissue thickness in predicting difficult airway risk in overweight and obese adult patients undergoing elective surgery under general anesthesia. Ultrasound-based anterior neck measurements will be compared with standard clinical airway assessment parameters to determine their diagnostic accuracy for difficult laryngoscopy and intubation.

The results of this study may contribute to improved preoperative airway risk stratification and safer airway management in obese patients.

DETAILED DESCRIPTION:
Difficult airway management remains a major concern in anesthetic practice and is associated with increased morbidity, particularly in obese patients. Excess anterior neck soft tissue and altered upper airway anatomy contribute to challenges in mask ventilation, laryngoscopy, and tracheal intubation. Conventional clinical airway assessment tests have limited predictive accuracy in this population, highlighting the need for additional objective assessment tools.

This prospective observational study is designed to evaluate the predictive value of ultrasound-based assessment of anterior neck soft tissue thickness for difficult airway risk in overweight and obese adult patients undergoing elective surgery under general anesthesia. The study will be conducted at a single tertiary care center after ethics committee approval, and written informed consent will be obtained from all participants.

Eligible patients aged 18-70 years with a body mass index (BMI) greater than 25 kg/m² and classified as ASA physical status I-III will be included. Emergency surgeries, pregnant patients, individuals with known difficult airway history, maxillofacial anomalies, neck masses, or a BMI greater than 60 kg/m² will be excluded.

Preoperative airway assessment will include conventional clinical parameters such as modified Mallampati score, mouth opening, interincisor distance, thyromental distance, sternomental distance, neck circumference, neck mobility, upper lip bite test, and snoring history. In addition, anterior neck ultrasound measurements will be performed preoperatively in the supine position using a high-frequency linear probe by trained anesthesiologists following a standardized protocol. Ultrasound parameters will include tongue dimensions, hyomental distance, skin-to-hyoid distance, skin-to-epiglottis distance, skin-to-vocal cords distance, skin-to-thyroid isthmus distance, skin-to-suprasternal notch distance, and the pre-epiglottic space to epiglottis-vocal cords distance ratio (PE/E-VC). Anterior neck ultrasound measurements will performed preoperatively by trained anesthesiologists using a standardized protocol.

A single prospective cohort of overweight/obese surgical patients will undergo preoperative ultrasound and clinical airway assessments, and outcomes during induction will be recorded. After induction of general anesthesia, laryngoscopic view will be assessed using the Cormack-Lehane classification. Difficult laryngoscopy will be defined as Cormack-Lehane grade III or IV. Intubation difficulty will be evaluated using the Intubation Difficulty Scale (IDS), and mask ventilation difficulty will be assessed using the Han scale. Intraoperative airway management data, including number of intubation attempts, need for adjuncts, alternative techniques, and airway-related complications, will be recorded.

Statistical analysis will focus on determining the diagnostic accuracy of ultrasound and clinical airway parameters. Receiver operating characteristic (ROC) curve analysis will be used to calculate the area under the curve (AUC), sensitivity, specificity, positive predictive value, and negative predictive value for each parameter and selected combinations. The findings aim to clarify the role of anterior neck ultrasound as a complementary tool for preoperative airway risk stratification in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* ASA physical status I-III

  * BMI >25 kg/m²
* Scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* Emergency surgery
* Pregnancy
* Maxillofacial anomalies or neck masses
* Rapid sequence induction
* Previous history of difficult intubation
* BMI >60 kg/m²

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overweight and obese adult patients undergoing elective surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Cormack-Lehane grade III-IV | During anesthesia induction
  Occurrence of difficult airway during anesthesia induction, defined by difficult laryngoscopy

SECONDARY OUTCOMES:
Ultrasound-derived anterior neck soft tissue measurements | During anesthesia induction
  diagnostic accuracy for predicting difficult airway (ROC-AUC)
Intubation Difficulty Scale (IDS) score | during tracheal intubation
  Difficult intubation: IDS score > 5
Han Scale | during ventilation
  Difficult mask ventilation: Han grade ≥ II

OTHER OUTCOMES:
Airway-related complications | during anesthesia induction
  Number of intubation attempts and need for airway adjuncts (stylet/bougie) and complications including desaturation and dental or soft tissue injury

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Nur Teke, medical doctor, Principal Investigator — Gaziantep City Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional data protection policies and the absence of participant consent for data sharing beyond the scope of the study.

REFERENCES:
- [Result] Udayakumar GS, Priya L, Narayanan V. Comparison of Ultrasound Parameters and Clinical Parameters in Airway Assessment for Prediction of Difficult Laryngoscopy and Intubation: An Observational Study. Cureus. 2023 Jul 5;15(7):e41392. doi: 10.7759/cureus.41392. eCollection 2023 Jul. PMID 37546081
- [Result] Kaul R, Singh D, Prakash J, Priye S, Kumar S, Bharati. Ultrasound Guided Measurement of Anterior Neck Tissue for the Prediction of Difficult Airway: A Prospective Observational Study. Rom J Anaesth Intensive Care. 2022 Dec 29;28(2):105-110. doi: 10.2478/rjaic-2021-0018. eCollection 2021 Dec. PMID 36844111
- [Result] Akin S, Yildirim M, Artas H, Bolat E. Predicting difficult airway in morbidly obese patients using ultrasound. Turk J Med Sci. 2023 Nov 21;54(1):262-274. doi: 10.55730/1300-0144.5787. eCollection 2024. PMID 38812631